CLINICAL TRIAL: NCT00204802
Title: A Patient-Centered Approach to Advance Care Planning of Patients With End Stage Heart Failure and Renal Disease
Brief Title: Patient-Centered Advance Care Planning
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2003-165
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2009-03

CONDITIONS: Heart Failure; Renal Failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

INTERVENTIONS:
Behavioral: Patient-Centered Advance Care Planning

SUMMARY:
Based on theories regarding decision-making and patient education the investigators have developed Patient-Centered Advance Care Planning (PC-ACP). This intervention is designed to improve patient and surrogate knowledge of ACP, increase the congruence between patient and surrogate in treatment decisions, decrease the patient's and surrogate's conflict in making such decisions, and increase the consistency between patient preferences and the actual care they receive. The ACP intervention is conducted with the patient in the presence of the surrogate.

ELIGIBILITY:
Inclusion Criteria:

* At high risk for impending death in the next 12 months

Exclusion Criteria:

* Patient not having decision-making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
efficacy of PC-ACP

CONTACTS AND LOCATIONS:
Overall Officials: Karin T Kirchhoff, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Kirchhoff KT, Hammes BJ, Kehl KA, Briggs LA, Brown RL. Effect of a disease-specific planning intervention on surrogate understanding of patient goals for future medical treatment. J Am Geriatr Soc. 2010 Jul;58(7):1233-40. doi: 10.1111/j.1532-5415.2010.02760.x. PMID 20649686